CLINICAL TRIAL: NCT03657108
Title: A Phase I Single-Arm Open Label Dose-Escalation Study of CivaSheet With Radical Prostatectomy With or Without Adjuvant External Beam Radiation Therapy in Patients With High Risk Prostate Cancer
Brief Title: CivaSheet With Radical Prostatectomy & Adjuvant External Beam Radiation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision made by DSMB to terminate study in April 2023.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ketan Badani, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1314; PD 16-03067 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-07-11; First posted 2018-09-04 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: brachytherapy; prostatectomy; radiation therapy; surgery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study to determine MTD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- group 1 of 60 Gy dose (Experimental): The first 3 subsequent patients with high risk prostate cancer will be undergoing radical prostatectomy Interventions: Civasheet 60 Gy + Adjuvant external beam radiation therapy
  Interventions: Radiation: Civasheet 60 Gy; Radiation: Adjuvant external beam radiation therapy
- group 2 of 60 Gy dose (Experimental): The second 3 subsequent patients with high risk prostate cancer will be undergoing radical prostatectomy Interventions: Civasheet 60 Gy + Adjuvant external beam radiation therapy
  Interventions: Radiation: Civasheet 60 Gy; Radiation: Adjuvant external beam radiation therapy
- group 1 of 75 Gy dose (Experimental): The third 3 subsequent patients with high risk prostate cancer will be undergoing radical prostatectomy Interventions: Civasheet 75 Gy + Adjuvant external beam radiation therapy
  Interventions: Radiation: Civasheet 75 Gy; Radiation: Adjuvant external beam radiation therapy
- group 2 of 75 Gy dose (Experimental): The fourth 3 subsequent patients with high risk prostate cancer will be undergoing radical prostatectomy Interventions: Civasheet 75 Gy + Adjuvant external beam radiation therapy
  Interventions: Radiation: Civasheet 75 Gy; Radiation: Adjuvant external beam radiation therapy

INTERVENTIONS:
Radiation: Civasheet 60 Gy — implantable proposed doses of Civasheet are 60 Gy
  Arms: group 1 of 60 Gy dose; group 2 of 60 Gy dose
Radiation: Civasheet 75 Gy — implantable proposed doses of Civasheet are 75 Gy
  Arms: group 1 of 75 Gy dose; group 2 of 75 Gy dose
Radiation: Adjuvant external beam radiation therapy — 45 Gy in 25 fractions
  Other Names: EBRT

SUMMARY:
A phase I single-arm open label dose escalation study to evaluate the maximum tolerated dose (MTD) and safety of Civasheet® with radical prostatectomy (RP) and adjuvant external beam radiation therapy (EBRT) in a 3+3 dose escalation design among participants with high risk prostate cancer (PCa).

DETAILED DESCRIPTION:
Using preoperative MRI imaging to identify areas suspicious of local advancement in addition to identifying areas with a higher likelihood of a positive margin during RP due to the presence of high risk features, Civasheet® and its inherently flexible structure allow the sheet to be directly implanted on areas suspicious for local advancement and positive surgical margins for direct application of radiation to these areas. The custom, single planar layer, integrative gold shielding of Civasheet® also allows radiation to be provided unidirectionally to allow healthy tissue (i.e., bladder, rectum) to be shielded from radiation; possibly affording a lower rate of gastrointestinal (GI) and genitourinary (GU) toxicity and adverse events. During EBRT, radiation especially for high risk PCa is provided at high rates to the entire prostatic bed with the seminal vesicles, pelvic lymph nodes and a surrounding margin often targeted to eliminate positive margins and cancer from locally advanced areas in which the cancer may have spread (i.e., seminal vesicles, bladder neck). These high rates of radiation often damage surrounding tissue and result in rectal and bladder complications in addition to urethral strictures among other adverse complications. Since Civasheet® will provide radiation to the prostatic bed, a lower dose of EBRT will be used to treat the prostatic bed and potentially lower adverse bladder and rectal effects compared to RP + RT at 60 Gy. 103 Pd seeds of Civasheet® also illuminate on imaging. Therefore placing Civasheet® based on pre-operative identification of areas suspicious for local advancement and areas of likely positive surgical margins during RP will allow for targeted EBRT to the locally advanced areas. Since EBRT can be targeted using Civasheet®, a lower and more direct dose of radiation during EBRT may be used to treat local advancement and positive surgical margins which will potentially reduce toxicity and complications associated with higher doses of radiation.

The above properties are likely to facilitate improved cancer control with more direct and local application of radiation to areas of local advancement surrounding the prostate. These features are also likely to facilitate a reduced complication and toxicity profile since Civasheet® allows EBRT to be applied more accurately and at a lower dose and also the unidirectional radiation applied directly by Civasheet® protects surrounding healthy tissue from receiving radiation.No other studies have attempted to use Civasheet® to improve PCa control and reduce toxicity and complications associated with radiation for participants with high-risk prostate cancer. The investigators anticipate that implanting Civasheet® on areas suspicious for local advancement and positive margins based on pre-operative MRI findings and identification of high risk features in addition to relying on the illumination provided by Civasheet® for targeted adjuvant EBRT will provide a safer complication profile and eventually provide evidence for superior cancer control, lower toxicity and less adverse events than EBRT+ RP alone in a future randomized controlled trial. The investigators therefore propose a phase I single-arm open label dose escalation study to evaluate the MTD and safety of Civasheet® with RP and adjuvant EBRT in a 3+3 dose escalation design among participants with high risk PCa.With this study, the investigators to better understand the MTD, safety and toxicity profile of Civasheet® in the setting of RP + adjuvant EBRT in the treatment of high-risk PCa.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with National Comprehensive Cancer Network (NCCN) very high or high risk adenocarcinoma of the prostate defined as ≥T3a, Gleason score ≥ 8, or PSA > 20 who is eligible for RP (open or robotic) with adjuvant EBRT as an initial treatment option.
* Any subject with NCCN Intermediate Risk adenocarcinoma of the prostate defined as T2b-T2c, Gleason score 7, or PSA 10-20 who is eligible for RP (open or robotic) with adjuvant EBRT as an initial treatment option and at least one of the following adverse features present in pre-operative imaging: seminal vesicle infiltration (SVI), extracapsular extension (ECE), N1 disease.
* Subject must have had a pre-operative MRI or must obtain a pre-operative MRI to be eligible for participation in this study.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Any subject who has undergone prior radiation to the pelvis.
* Subjects presenting with distant metastases.
* On any investigational drug(s), androgen deprivation therapy or therapeutic device(s) within 30 days preceding screening.
* Currently taking immunosuppressants, or with poorly controlled diabetes (HbA1c >8).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is a disease that only affects males. Therefore, this protocol will only recruit male patients with a prostate cancer diagnosis.
Enrollment: 6 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ketan K. Badani, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) sharing plan will be based on sharing patient information on REDcap. REDcap is an electronic database that will be used to share the data with other researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Duration of study
Access Criteria: Employed Mount Sinai Researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- 60 Gy: CivaSheet 60 Gy with fixed dose of adjuvant EBRT (45Gy)
- 75Gy: CivaSheet 75 Gy with fixed dose of adjuvant EBRT (45Gy)
Period: First Dose 60 Gy (90 Days Post EBRT)
Arm/Group | 60 Gy | 75Gy
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Next 2 Dose 60 Gy
Arm/Group | 60 Gy | 75Gy
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0
Period: First Dose 75 Gy (90 Days Post EBRT)
Arm/Group | 60 Gy | 75Gy
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Period: Next 2 Dose 75 Gy
Arm/Group | 60 Gy | 75Gy
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 Gy | 75Gy | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 56 [55 to 61] | 56 [53 to 71] | 56 [53 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 0 | 2 | 2
  Non-Hispanic Black | 1 | 1 | 2
  Hispanic | 2 | 0 | 2
American Society of Anesthesiologists score (ASA) [Count of Participants; unit: Participants] — ASA I: A normal healthy patient.
  ASA II: A patient with mild systemic disease.
  ASA III: A patient with a severe systemic disease that is not life-threatening.
  Participants
    I | 1 | 0 | 1
    II | 1 | 3 | 4
    III | 1 | 0 | 1
Magnetic Resonance Image (MRI) Tumor size [Median (Full Range); unit: cm] | 3 [2.3 to 5.3] | 1.5 [1.5 to 5.3] | 2.7 [1.5 to 5.3]
MRI extracapsular extension [Count of Participants; unit: Participants] | 2 | 0 | 2
MRI seminal vesicle infiltration [Count of Participants; unit: Participants] | 1 | 0 | 1
MRI nodal disease [Count of Participants; unit: Participants] | 1 | 0 | 1
MRI metastasis [Count of Participants; unit: Participants] | 0 | 0 | 0
Baseline Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 26.3 [8.3 to 43.8] | 38.6 [5.1 to 41.5] | 32.5 [5.1 to 43.8]
Biopsy grade group [Count of Participants; unit: Participants] — Grade 1 - The cancer is likely to grow and spread very slowly (called well differentiated or low grade).
  Grades 2 - The cancer is likely to grow and spread slowly (called moderately differentiated or intermediate grade).
  Grades 3 - The cancer is more likely to grow and spread than Grade Group 2 (called moderately differentiated or intermediate grade).
  Grades 4 - The cancer is likely to grow and spread quickly (called poorly differentiated or high grade).
  Grade 5 - The cancer is likely to grow and spread more quickly than Grade Group 4 (called poorly differentiated or high grade).
  Participants
    1 | 0 | 0 | 0
    2 | 1 | 1 | 2
    3 | 1 | 1 | 2
    4 | 1 | 0 | 1
    5 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerable Dose (MTD)
Description: MTD is defined as the highest dose of the Civasheet® not yielding unacceptable toxicity. Specifically if > 33 % of subjects experience dose limiting toxicity (DLT) at any dose level, the dose level below that level will be considered the MTD.
Time Frame: 90 days
Measure: Number; unit: Gy
Groups:
- All Participants: All participants who received at least 1 dose of CivaSheet, either at 60 Gy or 75 Gy with fixed dose of adjuvant external beam radiation therapy (EBRT) (45Gy)
Arm/Group | All Participants
Number analyzed (Participants) | 6
Gy | 75

2. Secondary Outcome: Number of Surgical Complications
Description: Number of surgical major complications (major complications defined as Clavien≥3.):
  intraoperative, post operative - acute (< 90 days) and late (18 months).
  Grade III - Requiring surgical, endoscopic or radiological intervention
  Grade IV - Life-threatening complication (including central nervous system (CNS) complications) requiring intensive care (IC/ICU)-management
  Grade V - Death of a patient
Time Frame: intraoperative, postoperative - acute (< 90 days) and late (18 months)
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants
  Intraoperative complication | 0 | 0
  Postoperative complication | 0 | 0
  intraoperative, postoperative - acute (< 90 days) and late (18 months) | 0 | 0

3. Secondary Outcome: Number of Participants With Biochemical Recurrence (BCR)
Description: Number of participants with Biochemical recurrence (BCR) at 6-month follow-up after EBRT. BCR was defined as a post-prostatectomy serum prostate-specific antigen (PSA) level greater than 0.2 nanograms per milliliter (ng/mL).
Time Frame: 6-month follow-up after EBRT
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With Erectile Dysfunction
Description: Number of participants with Erectile Dysfunction at least 6 months after EBRT
Time Frame: 6 months after EBRT
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants | 3 | 2

5. Secondary Outcome: Number of Participants With PSA Persistence
Description: Number of participants with PSA persistence which is defined as PSA persistently greater than 0.2 ng/mL after surgery.
Time Frame: 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With Urinary Incontinence
Description: Number of Participants with Urinary Incontinence at least 6 months after EBRT
Time Frame: at least 6 months after EBRT, up to 40 months
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Acute Radiation Toxicity
Description: Number of participants with Acute (occurring within 90 days) radiation toxicity using the Radiation Therapy Oncology Group (RTOG) Acute Toxicity Scale and Late Radiation Morbidity scales; including Grade 4-5 hematuria, fistula formation, proctitis or death.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants | 0 | 1

8. Other Pre Specified Outcome: Number of Participants With Late Radiation Toxicity
Description: Number of participants with Late (occurring after 90 days) radiation toxicity using the Radiation Therapy Oncology Group (RTOG) Acute Toxicity Scale and Late Radiation Morbidity scales; including Grade 4-5 hematuria, fistula formation, proctitis or death.
Time Frame: after 90 days, up to 4 years 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

9. Other Pre Specified Outcome: Number of Radiation Adverse Event(s)
Description: National Cancer Institute's Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v4.0); 5 Grades where Grade 1 is the better outcome and Grade 5 is the worse outcome
Time Frame: 4 years 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | 60 Gy | 75Gy
Number analyzed (Participants) | 3 | 3
Participants
  Grade 1 - Mild Adverse Event | 0 | 1
  Grade 2 - Moderate Adverse Event | 0 | 0
  Grade 3 - Serious Adverse Event | 0 | 0
  Grade 4 - Life-threatening Adverse Event | 0 | 0
  Grade 5 - Fatal Adverse Event | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years, 10 months for participants who received EBRT 1 year for participants who did not receive EBRT
Arm/Group | 60 Gy | 75Gy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 Gy (N=3) | 75Gy (N=3)
Radiation cystitis (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03657108/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03657108/SAP_001.pdf
  • Informed Consent Form (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03657108/ICF_002.pdf